CLINICAL TRIAL: NCT00319358
Title: Effect of Antioxidant Supplementation on Pain, Antioxidant Profile and Oxidative Stress in Patients With Chronic Pancreatitis
Brief Title: Role of Antioxidants Supplementation in Chronic Pancreatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR-131
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Pancreatitis
Keywords: chronic pancreatitis; antioxidant supplementation; oxidative stress
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Antioxidants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antioxidants (Active Comparator): Intervention was done with antioxidants
  Interventions: Dietary Supplement: Antioxidants
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Antioxidants — 600microgm selenium, 0.54g vitamin C, 9000IU beta-carotene, 270IU vitamin E, 2g methionine per day, daily, in divided doses for 6 months
  Other Names: Betamore G, Osper Pharmanautics, India
  Arms: Antioxidants
Dietary Supplement: Placebo — placebo
  Arms: Placebo

SUMMARY:
Chronic pancreatitis is a progressive inflammatory disease of the pancreas that presents with abdominal pain and in late stages may cause diabetes and malnutrition. The pain may be incapacitating and may affect patients physically, mentally and socially. Pain due to chronic pancreatitis is difficult to treat. Oxidative stress and free radical mediated injury has been shown to cause pancreatic inflammation. It has been shown that patients with chronic pancreatitis are deficient in micronutrients and natural antioxidants such as b-carotene, vitamin E and C etc. Studies have suggested that antioxidant supplementation may help to combat pain in these patients. Antioxidant supplementation may decrease the oxidative stress and boost the antioxidant status, thereby resulting in pain relief. The investigators have planned to perform a trial to study the effect of antioxidant supplementation on pain relief in patients with chronic pancreatitis.

DETAILED DESCRIPTION:
INTRODUCTION Chronic pancreatitis (CP) is a progressive inflammatory disease of the pancreas accompanied by abdominal pain and in late stages, by exocrine and endocrine insufficiency. The etiology of CP include alcohol abuse, hereditary, ductal obstruction, tropical pancreatitis, systemic diseases (systemic lupus erythematosus and cystic fibrosis etc.), and idiopathic. Alcohol abuse accounts for 70-80% of cases of chronic pancreatitis in the West and about 40% in India. The intensity of injury depends on the duration and amount of alcohol consumed. Hereditary pancreatitis transmitted as an autosomal dominant trait accounts for a small subset of all cases of CP, and occurs due to mutation in cationic trypsinogen gene. Pancreatic duct obstruction may be secondary to trauma, pseudocysts, calcific stones or tumors and leads to obstructive CP (1). Tropical pancreatitis is a condition of unknown etiology that is seen predominantly in south India and other tropical areas of the World. Young patients are commonly affected with this disease. Cassava consumption had been proposed as an etiological factor due to its cyanogenic glycoside content however no epidemiological study has proved this hypothesis (2). Malnutrition has been suggested as an etiological factor in tropical pancreatitis. Idiopathic pancreatitis accounts for a substantial number of cases.

Many recent studies have emphasized a role for Reactive Oxygen Radicals (ROR) in the development of oxidative stress and hence inflammation in the pathogenesis of chronic pancreatitis. Increased oxidative stress probably results from increased exposure to xenobiotics. Xenobiotics are chemical substances present in the environment to which human beings are constantly exposed. It is conceivable that many of these xenobiotics are metabolized in pancreas that contains cytochrome P450 (CYP450) enzymatic system. The metabolism of xenobiotics occurs through two phases, Phase I and Phase II. Phase I metabolism may result in 'bioactivation' of the xenobiotics, in turn activating CYP system. Phase II involves attachment of biotransformed compound to a biological molecule that makes it more polar and thus easier to excrete. The metabolism of xenobiotics places an oxidative stress and can overwhelm the natural antioxidant defense of the body. The resultant production of the free radicals may play an important role in the pathogenesis of CP (2). Over induction of this enzyme can cause increased utilization of glutathione (GSH), which causes irreversible loss of glutathione. Moreover glutathione serves as a reservoir for cysteine/cystine required for disulphide synthesis for pancreatic digestive proteins. This further aggravates the situation. Three types of cytochrome enzymes are induced through xenobiotics. CYP2E1 has been specifically examined in the context of liver injury. CYP1A metabolizes smoke constituents and potent carcinogens such as benzo(a)pyrene. Cytochrome 3A is inducible by reactive oxygen species generated from aflatoxin B1. Alcohol, nicotine from cigarette smoke and other forms of tobacco consumption and industrial pollutants all are considered as xenobiotics and overwhelm the detoxification capacity of cytochrome CYP450 system (3). The CYP induction increases heme and heme-oxygenase thus buttressing the antioxidant defenses. The free radical peroxidation products may act as second messengers and block exocytosis leading to increased autophagy and crinophagy thus diverting the pancreatic enzymes into interstitium. This leads to degranulation of mast cells inducing inflammation mediated by chemotaxis. The synthesis of enzyme proteins in pancreas also produces H2O2, which also induces free radical production. Furthermore the depressed methionine trans-sulphuration pathway induces CYP as well. The free radicals generated from all these processes induce oxidative stress, which is implicated in damage to cell membranes due to lipid peroxidation. Above all, if the antioxidant levels of an individual are may be low due to either low intake or depletion during oxidative stress. Some studies also indicate that free radicals cause disintegration of antioxidative enzymes if over exposed to them.

However, the role of oxidative stress still not fully explained in that whether the oxidative stress is the cause of chronic pancreatitis or a consequence of it. This can be established by two observations: 1) If the oxidative stress is noted before the onset of disease and 2) If the disease symptoms are relieved by supplementation with antioxidants. Patients with alcoholic pancreatitis have been shown to have an increased oxidative stress. Supplementation with antioxidants hence decreases the production of such free radicals and may be beneficial to patients with CP (4).

A study by Braganza et al has shown that CP involves oxidative stress in-patients with CP (5). This was the first study to indicate the role of free radicals in the pathogenesis of chronic pancreatitis. However, the mechanism by which it occurs is still unclear. The preliminary studies show that malondialdehyde (MDA); a marker of peroxidation secondary to oxidative stress increases during CP.

In the present proposed study, the aim is to find out if there is increased oxidative stress in patients with CP and if supplementation with antioxidants relieves pain in them in order to establish a relationship between oxidant stress and pathophysiology of chronic pancreatitis.

Objectives

1. To evaluate the effect of antioxidant supplementation given daily on pain relief in chronic pancreatitis during the 6 months of therapy as compared to a placebo.
2. To assess the improvement in oxidative stress and antioxidant profile in these patients during 6 months of antioxidant supplementation by measuring markers of oxidative stress and blood antioxidant levels.

Material and methods Study Design: Double blind randomized controlled trial Patients All consecutive patients with chronic pancreatitis attending the pancreas clinic at AIIMS will be included in the study as per the inclusion criteria. The diagnosis of CP will be made if there is evidence of CP on imaging studies including plain film of the abdomen, Ultrasonography, Computerized tomography (CT) scan, endoscopic retrograde cholangiopancreatography (ERCP), and magnetic resonance imaging (MRI) scan. Also hematological tests, biochemical investigations will be done as part of diagnostic work-up.

All patients will undergo detailed clinical evaluation including detailed family history of pancreatic diseases and diabetes. The WHO criteria will be used to diagnose diabetes. The patients will also be inquired about their dietary history and addiction to tobacco or alcohol. Patients will be explained the purpose of study clearly and consent forms will be duly signed by them. The patients will be regularly followed up in pancreas clinic at All India Institute of Medical Sciences, New Delhi. All the patients will be treated in the standard manner including medical, endoscopic and surgical treatment as and when indicated.

Inclusion criteria:

CP with significant pain i.e. at least one episode of pain in a month requiring oral analgesic or one episode of severe pain in last three months requiring hospitalization.

Sample size calculation Sample size is calculated on the basis of probability sampling methods. For 80% power at a significance level of 5% (a = 0.05), a sample size of 100 in each arm would be required.

Randomization and blinding Randomization of treatment allocation largely ensures unbiased treatment comparison. A simple randomization scheme for treatment allocation will be done using a table of random numbers by a Statistician/ Epidemiologist not associated with conduct of the study. He/she will label the boxes of treatment with individual patient numbers from 1-200 according to the randomization scheme. This person will keep the assignment code at a safe place; the code will be available to the investigator only at the end of the trial. These will be serially opened as new patients are recruited into the study. Double blinding will be done to ensure minimum bias i.e. blinding of researcher and clinician attending patients to the randomization process so that allocation and outcome evaluation are not affected and blinding of patients to the identity of the drug or intervention they are receiving. The inert placebo, which will be identical to the active drug in packaging, appearance and schedule of administration.

Intervention One group will be given antioxidant supplementation and the other group will be placebo. The antioxidant intervention will be daily doses of 600 mg organic selenium, 0.54 g vitamin C, 9000 IU B-carotene, 270 IU vitamin E and 2 g methionine. Both the groups will be supplemented with the pancreatic enzymes. The enzyme will be administered as capsules, each containing 10,000 units. Three capsules (30,000) units will be required per meal thereby making it to 90,000 units per day.

Follow up assessment during study period:

Clinical:

* Assessment of painful days and requirement of oral/ IV analgesic or hospitalization in a month will be done. The patients will be provided with a pain diary so as to get the correct data.
* Any other symptoms either due to primary disease i.e. CP or considered due to the intervention will be duly recorded.

  * Pain assessment and clinical examination will be done at each visit of patient to the clinic while USG, ERCP, CT or X-ray will be done as and when required.

Markers of oxidative stress

* MDA Marker of antioxidant capacity or defense
* Superoxide dismutase (SOD), Total glutathione, Ferric Reducing Assay of Plasma (FRAP) Markers of intervention compliance
* Vitamins A, E, C *All the biochemical investigations will be done at baseline, 1 and 6 months of intervention.

All the samples will be light protected and purged with nitrogen to retard deterioration from oxidation of substrates during storage.

Statistics Descriptive statistics i.e. mean, standard deviation and frequency distribution will be calculated for each variable in the study. To compare the two groups, Student 't' test (quantitative) and chi square test (qualitative) wherever applicable will be applied. To see trend within the variable 2-way analysis of variance (parametric as well as non-parametric, whichever is applicable) will be done post-hoc analysis. P value < 0.05 will be considered as statistical significant. Statistic software SPSS 7.5 for Windows will be used for statistical analysis.

Study Outcome Primary Outcome

1. Reduction in the number of painful days per month due to chronic pancreatitis.

Secondary Outcome

1. Decrease in no. of severe attacks requiring hospitalization.
2. Percentage of patients who are pain-free.
3. Increase in markers of antioxidant defense in the intervention group compared to placebo group and decrease in oxidative stress parameters in patients after intervention compared to placebo.

References:

1. Pitchumoni CS, Mohan AT. Pancreatic stones. Gastroenterol. Clin. North Amer. 1990: 19; 873-893.
2. Walling MA. Xenobiotic metabolism, oxidant stress and chronic pancreatitis: Focus on glutathione. Digestion 59 (Suppl4): 13-24, 1998.
3. Lin Y, Tamakoshi A et al. 2000. Cigarette smoke as a risk factor for chronic pancreatitis: A case control study in Japan. Pancreas. 21 (2), 109-114.
4. Uden S, Schofield D, Miller PF, Day JP Bottiglier T and Braganza JM. 1992. Aliment Pharmacol Ther. 6, 229-240.
5. Braganza JM. A framework for etiogenesis of chronic pancreatitis. Digestion: 1998; 59 (suppl. 4): 1-12.

ELIGIBILITY:
Inclusion Criteria:

* CP with significant pain i.e., at least one episode of pain in a month requiring oral analgesic or one episode of severe pain in last three months requiring hospitalization

Exclusion Criteria:

* Painless disease
* Current pain more likely due to non-pancreatic origin
* If the patient already has an intervention in the form decompressive therapy i.e., surgery or endoscopic sphincterotomy/ stenting or ESWL
* Systemic conditions like CRF, malignancy, hypertension, and pregnancy
* Complications like pseudocyst, pancreatic abscess
* Patients who would have received antioxidants in the preceding 4 weeks
* Narcotic addicts
* Uncontrolled diabetes
* Comorbid conditions like liver diseases

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2003-10; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Reduction in the number of painful days per month due to chronic pancreatitis | 6 months

SECONDARY OUTCOMES:
Decrease in no. of severe attacks requiring hospitalization | 6 months
Percentage of patients who are pain-free | 6 months
Increase in markers of antioxidant defense in the intervention group compared to placebo group and decrease in oxidative stress parameters in patients after intervention compared to placebo | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Payal Bhardwaj, MSc, Principal Investigator — dept. of Gastroenterology, A.I.I.M.S. , New Delhi; Pramod K Garg, MD, DM, Study Director — Dept. of Gastroenterology, All India Institute of Medical Sciences, New Delhi
Locations (1):
- A.I.I.M.S., New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Chouduary A, Garg PK, Tandon RK. The role of oxidative stress in tropical pancreatitis and effect of antioxidants supplementation on pain in patients with tropical pancreatitis. J Gastroenterol. Hepatol. 2001;16(Suppl):A132(Abstract).
- [Background] McCloy R. Chronic pancreatitis at Manchester, UK. Focus on antioxidant therapy. Digestion. 1998;59 Suppl 4:36-48. doi: 10.1159/000051441. PMID 9832634